CLINICAL TRIAL: NCT04870450
Title: When Distance is an Act of Love: Exploring the Use of Video Diaries for Family Members of Intensive Care Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government); University of Hertfordshire (Other)
Responsible Party: Principal Investigator, Sheila Rodgers, Senior Lecturer, University of Edinburgh
Other Study IDs: CAHSS2010/07
Record Dates: First submitted 2021-01-25; First posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Coronavirus; Anxiety Depression
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthcare professionals: No intervention. Gathering data on their experiences of using video diaries.
- Family members of ICU patients: No intervention. Gathering data on their experiences of using video diaries.

SUMMARY:
Due to Covid-19, intensive care (ICU) patients are not allowed visitors or have severely restricted visiting. After being admitted to ICU most patients are unconscious or extremely weak and therefore cannot speak on a phone or video call to a family member. Before these visiting restrictions, family members of patients admitted to ICU as a result of being critically ill were already known to suffer significant psychological distress and may now face increased distress given they are unable to visit a loved one.

Previous research demonstrates that keeping a paper diary has been found to be helpful for ICU patients and families. When lockdown measures were announced, NHS Scotland introduced video diaries as an emergency measure to try to support communication with families and reduce distress. vCreate is an NHS Trusted secure video messaging service that helps patients, families and clinical teams stay connected throughout their care journey. The use of video diaries may have a positive impact for family members but there is a risk that they could also have negative effects for some people. There is a need to explore both ICU healthcare professionals and family members' experiences of using video diaries. At the same time it is also important to test the feasibility and acceptability of measures of distress and psychological well-being on family members during and after their experience of video diaries. In doing so, some initial recommendations about video diaries can be made and a larger subsequent study planned to test their effect on family members and healthcare professionals.

ELIGIBILITY:
Inclusion Criteria:

- (i) Family Members in Lothian aged ≥16 years receiving a video diary for an ICU patient who stays in ICU for ≥24 hours or more. If the patient dies, family members will be invited to continue in the study.

(ii) ICU healthcare staff in NHS Lothian who have experience of using the video diary to support family members during lockdown.

Exclusion Criteria:

Prisoners Family members lacking capacity to consent Family members aged under 16 years

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We aim to recruit up to 20 family members who were involved with using video diaries and up to 8 healthcare professionals who supported family members of ICU patients through video diaries. We will recruit family members and healthcare professionals from two of NHS Lothian's ICU's.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2021-01-26 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Qualitative experiences | 3 months
  The principal aim of this study is to explore the experiences of family members and healthcare professionals in using video diaries during the lockdown and no/very restricted hospital visiting.

SECONDARY OUTCOMES:
WEMWBS | 3 months
  (Warwick-Edinburgh Mental Well-being Scale) is a tool that measures psychological well-being.
CORE-OM | 3 months
  CORE-OM (Clinical Outcomes in Routine Evaluation-Outcome Measure) is a self report of a non-proprietary, pan-theoretical (not allied to any particular modality) measure of global psychological distress.
Daily Distress Thermometer | 3 months
  The Daily Distress thermometer is an adaptation of the National Comprehensive Cancer Network Distress Thermometer and Problem list.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Edinburgh, Edinburgh, Lothian, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gazzato A, Scquizzato T, Imbriaco G, Negro A, Caballo Garrido MC, Landoni G, Zangrillo A, Borghi G. The Effect of Intensive Care Unit Diaries on Posttraumatic Stress Disorder, Anxiety, and Depression: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Dimens Crit Care Nurs. 2022 Sep-Oct 01;41(5):256-263. doi: 10.1097/DCC.0000000000000539. PMID 35905428